CLINICAL TRIAL: NCT01229956
Title: Promoter Methylation in MLL-Rearranged Childhood AML
Brief Title: Biomarkers in Tissue Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B3; COG-AAML11B3 (Other: Children's Oncology Group); NCI-2011-02842 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B3 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer the in laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether the pattern of global and TSG-specific promoter CpG island hypermethylation and gene silencing that we have shown characterizes MLL-rearranged (MLL-r) infant bilineage ALL is also characteristic of other subsets of MLL-r leukemia.

OUTLINE: Previously collected cryopreserved cells from diagnosis are analyzed for promoter methylation via HELP arrays, gene expression arrays, and RT-qPCR.

PROJECTED ACCRUAL: A total of 32 samples (8 from each of 4 biologically defined cohorts) will be analyzed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Available cryopreserved cells from diagnosis

  * At least 2 x 10^7 viably cryopreserved cells
* One of the following biologically defined cytogenetics/molecular cohorts:

  * t(9;11)
  * t(11;19)
  * Other 11q23 translocations
  * Normal cytogenetics

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients With Acute Myeloid Leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of differential patterns of promoter hypermethylation and gene expression in pairwise comparisons with other cohorts and normal controls

CONTACTS AND LOCATIONS:
Overall Officials: Patrick N. Brown, MD, Principal Investigator — CHRISTUS Santa Rosa Cancer Center at CHRISTUS Santa Rosa Hospital - City Centre